CLINICAL TRIAL: NCT01536418
Title: A Randomised, Double-blind, Active Treatment Study to Induce Clinical Response and/or Remission With GSK1605786A in Subjects With Moderately-to-Severely Active Crohn's Disease
Brief Title: An Active Treatment Study to Induce Clinical Response and/or Remission With GSK1605786A in Subjects With Crohn's Disease
Acronym: SHIELD-4
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 114643
Record Dates: First submitted 2012-02-16; First posted 2012-02-22 (Estimated); Results first posted 2017-08-17 (Actual); Last update posted 2018-01-29 (Actual); Status verified 2018-01

CONDITIONS: Crohn's Disease
Keywords: Crohn's disease, chemokine receptor 9 antagonist, Crohn's Disease Activity Index; active treatment
MeSH Terms: conditions — Crohn Disease | interventions — CCX282-B

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- GSK1605786A, 500 milligrams, once daily (Experimental): 500 milligrams once daily, orally administered for 12 weeks
  Interventions: Drug: GSK1605786A
- GSK1605786A, 500 milligrams twice daily (Experimental): 500 milligrams twice daily, orally administered for 12 weeks
  Interventions: Drug: GSK1605786A

INTERVENTIONS:
Drug: GSK1605786A — 500 milligrams once daily, orally administered for 12 weeks
  Arms: GSK1605786A, 500 milligrams, once daily
Drug: GSK1605786A — 500 milligrams twice daily, orally adminstered for 12 weeks
  Arms: GSK1605786A, 500 milligrams twice daily

SUMMARY:
This is a multi-centre, randomised, double-blind, active treatment, parallel group induction study in subjects with moderately-to-severely active Crohn's disease. Subjects will receive one of two doses (500 milligrams once daily, 500 milligrams twice daily) of GSK1605786A for 12 weeks. The primary objective of the study is to induce clinical response (Crohn's Disease Activity Index [CDAI] decrease from baseline of at least 100 points) and/or remission (CDAI score less than 150) with GSK1605786A at Week 12 in subjects with active Crohn's disease to qualify subjects for enrolment into a 52 week maintenance study (CCX114157). Secondary objectives will include assessment of the safety and evaluation of the efficacy in induction of clinical response or remission. Safety will be assessed by recording of adverse events and assessment of changes in clinical laboratory parameters, vital signs and electrocardiogram. Population pharmacokinetics will evaluate the two doses of GSK1605786A. Health outcomes assessments will include changes in Inflammatory Bowel Disease Questionnaire, SF-36, EQ-5D, and Work Productivity and Activity Impairment-Crohn's Disease.

DETAILED DESCRIPTION:
This is a multi-centre, double-blind, randomised, active treatment, parallel group study designed to induce clinical response and/or clinical remission with two oral doses of GSK1605786A (500 milligrams once daily, 500 milligrams twice daily) over a 12-week treatment period in subjects with moderately-to-severely active Crohn's disease. The primary objective of this study is to qualify subjects for enrolment into a follow up 52 week maintenance study CCX114157. Subjects who achieve induction of clinical response (CDAI decrease from baseline of at least 100 points) or remission (CDAI score less than 150) at Week 12 following treatment with GSK1605786A will be eligible for enrolment into the maintenance study CCX114157. Secondary objectives will include assessment of the safety and evaluation of the efficacy in induction of clinical response or remission.

The study is planned to randomise approximately 900 subjects (450 subjects per group) with active Crohn's disease who have been diagnosed for at least 4 months, with documented history of disease in the small and/or large intestine, and characterised by a CDAI score between 220 to 450 (inclusive). Subjects will be required to have evidence of current active inflammation by elevated C-reactive protein (greater than the upper limit of normal of the highly sensitive C-reactive protein test) OR an elevated level of faecal calprotectin. Subjects will be allowed to participate in the study while continuing on stable doses of agents typically used to treat Crohn's disease. Inclusion of subjects who received prior treatment with an anti-tumor necrosis factor agent and discontinued due to loss or lack of efficacy will be limited to approximately 50 percent of the study population. Following a 3-week screening period, subjects will be randomised at baseline to receive blinded treatment with one of two doses of GSK1605786A (500 milligrams once daily or twice daily) for 12 weeks. All subjects meeting the definition of responder (CDAI decrease from baseline of at least 100 points) or who are in remission (CDAI score less than 150 points) at Week 12 will be eligible for randomisation into an ongoing maintenance study (CCX114157). Subjects who do not meet the definition of responder or who are not in remission at Week 12 will not be eligible to participate in study CCX114157.

For subjects who complete the study the minimum duration of participation is 15 weeks and the maximum duration is 19 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects aged 18 years or older
* Written informed consent prior to any of the screening procedures including discontinuation of prohibited medications
* Diagnosis of Crohn's disease for more than 4 months with small bowel and/or colonic involvement
* Current evidence of moderately-to-severely active disease defined by a baseline Crohn's Disease Activity Index (CDAI) score of 220 to 450, inclusive
* Confirmation of active disease by elevated CRP (greater than or equal to the upper limit of normal for the highly sensitive C-reactive protein test) or elevated levels of faecal calprotectin
* History of inadequate response and/or intolerance or adverse event leading to discontinuation of at least one of the following treatments for Crohn's disease: corticosteroids or immunosuppressants
* Stable doses of permitted concomitant medications or having previously received, but are not currently receiving, medications for Crohn's disease
* Demonstrated ability to comply with Crohn's disease symptom recording using the interactive voice response system
* Female subjects of child-bearing potential are eligible if not pregnant or nursing and committed to use of contraceptive methods with a failure rate of less than 1 percent per year

Exclusion Criteria:

* Known coeliac disease, those who follow a gluten-free diet to manage symptoms of suspected coeliac disease and subjects with a positive screening test for coeliac disease (elevated anti-tissue transglutaminase antibodies)
* Diagnosis of ulcerative or indeterminate colitis
* Enterocutaneous, abdominal or pelvic fistulae with abscesses, or fistulae likely to require surgery during the course of the study period
* Bowel surgery, other than appendectomy, within 12 weeks prior to screening and/or has planned surgery or deemed likely to need surgery for Crohn's disease during the study period
* Extensive colonic resection, subtotal or total colectomy
* Presence of ileostomies, colostomies or rectal pouches
* Fixed symptomatic stenoses of small bowel or colon
* History of more than 3 small bowel resections or diagnosis of short bowel syndrome
* Chronic use of narcotics for chronic pain defined as daily use of one or more doses of narcotic containing medicaitons
* Use of prohibited medications, including enteral feeding or elemental diet, within their specified timeframes and throughout the study. Prohibited medications include the following:

  1. Biologic use: Use of any TNF inhibitor (such as infliximab, adalimumab or certolizumab) or natalizumab within 10 weeks prior to Randomisation
  2. Corticosteroid use: Use of parenteral glucocorticoids within 4 weeks prior to Screening
  3. Immunospressant use: Use of cyclosporine, tacrolimus, sirolimus or mycophenolate mofetil within 4 weeks prior to Screening
  4. Intravenous antibiotic use: Use of intravenous antibiotics for Crohn's disease within 4 weeks prior to Screening
  5. Enteral feeding: Use of tube or enteral feeding, elemental diet within 2 weeks prior to Screening
  6. Rectal Treatment: Use of 5-aminosalicylates or corticosteroid enemas or suppositories within 2 weeks prior to Screening
  7. Leukocytapheresis or granulocytapheresis within 2 weeks prior to Screening
  8. Paracetamol or acetaminophen greater than 2 grams per day
  9. Opioid analgesics for worsening Crohn's disease pain are prohibited when used on a regular daily basis for more than 3 days
  10. Digoxin or related cardiac glycosides: Use within 7 days prior to Screening
  11. Any previous participation in a clinical study of GSK1605786A (formerly ChemoCentryx compound CCX282-B)
* Positive immunoassay for Clostridium difficile
* Known HIV infection
* Known varicella, herpes zoster, or other severe viral infection within 6 weeks of screening
* Immunization with a live vaccine within 4 weeks of Screening and throughout the study with the exception of the influenza vaccine
* Positive hepatitis B surface antigen or hepatitis B core antibody test or positive Hepatitis C test result at Screening
* Active or latent tuberculosis infection determined by results of QuantiFERON TB Gold test
* Current sepsis or infections requiring intravenous antibiotic therapy for more than 2 weeks
* Previous infections characterised by opportunistic pathogens, and/or dissemination suggestive of clinically significant immunocompromise
* Evidence of hepatic dysfunction, viral hepatitis, or abnormalities in liver function test results
* Corrected QT interval of ECG (electrocardiogram) greater than or equal to 450 milliseconds
* Congenital or acquired immunodeficiency or has evidence of immunocompromise manifested by current opportunistic infection
* Current evidence of, or has been treated for a malignancy within the past five years (other than localised basal cell, squamous cell skin cancer, cervical dysplasia, or any cancer in situ that has been resected)
* History of evidence of adenomatous colonic polyps that have not been removed.
* History of evidence of colonic mucosal dysplasia
* If female, is pregnant, has a positive pregnancy test or is breast-feeding
* Concurrent illness or disability that may affect the interpretation of clinical data, or otherwise contraindicates participation in this clinical study (such as an unstable cardiovascular, autoimmune, renal, hepatic, pulmonary, endocrine, metabolic, gastrointestinal, haematologic, or neurological condition or mental impairment)
* Medical history of sensitivity to any of the components of GSK1605786A (microcrystalline cellulose, crospovidone, sodium stearyl fumarate).
* Use of any investigational product within 30 days prior to screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 255 (Actual)
Dates: Start 2011-11-11 (Actual); Primary Completion 2013-10-17 (Actual); Study Completion 2013-10-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (192):
- United States (38):
  - GSK Investigational Site, Little Rock, Arizona
  - GSK Investigational Site, Tucson, Arizona
  - GSK Investigational Site, La Jolla, California
  - GSK Investigational Site, Aurora, Colorado
  - GSK Investigational Site, Denver, Colorado
  - GSK Investigational Site, Littleton, Colorado
  - GSK Investigational Site, Hamden, Connecticut
  - GSK Investigational Site, New Haven, Connecticut
  - GSK Investigational Site, Washington D.C., District of Columbia
  - GSK Investigational Site, Jacksonville, Florida
  - GSK Investigational Site, Port Orange, Florida
  - GSK Investigational Site, Suwanee, Georgia
  - GSK Investigational Site, Chicago, Illinois
  - GSK Investigational Site, Chevy Chase, Maryland
  - GSK Investigational Site, Towson, Maryland
  - GSK Investigational Site, Boston, Massachusetts
  - GSK Investigational Site, Chesterfield, Michigan
  - GSK Investigational Site, Rochester, Minnesota
  - GSK Investigational Site, Lee's Summit, Missouri
  - GSK Investigational Site, Mexico, Missouri
  - GSK Investigational Site, Brooklyn, New York
  - GSK Investigational Site, Lake Success, New York
  - GSK Investigational Site, Stony Brook, New York
  - GSK Investigational Site, Chapel Hill, North Carolina
  - GSK Investigational Site, Charlotte, North Carolina
  - GSK Investigational Site, Columbus, Ohio
  - GSK Investigational Site, Tulsa, Oklahoma
  - GSK Investigational Site, Portland, Oregon
  - GSK Investigational Site, Pittsburgh, Pennsylvania
  - GSK Investigational Site, Nashville, Tennessee
  - GSK Investigational Site, Austin, Texas
  - GSK Investigational Site, Ogden, Utah
  - GSK Investigational Site, Christiansburg, Virginia
  - GSK Investigational Site, Danville, Virginia
  - GSK Investigational Site, Norfolk, Virginia
  - GSK Investigational Site, Richmond, Virginia
  - GSK Investigational Site, Madison, Wisconsin
  - GSK Investigational Site, Milwaukee, Wisconsin
- Australia (6):
  - GSK Investigational Site, Bankstown, New South Wales
  - GSK Investigational Site, Adelaide, South Australia
  - GSK Investigational Site, Box Hill, Victoria
  - GSK Investigational Site, Fitzroy, Victoria
  - GSK Investigational Site, Prahran, Victoria
  - GSK Investigational Site, Fremantle, Western Australia
- Austria (5):
  - GSK Investigational Site, Hall in Tirol
  - GSK Investigational Site, Linz
  - GSK Investigational Site, Oberpullendorf
  - GSK Investigational Site, St.Veit/Glan
  - GSK Investigational Site, Vienna
- Belgium (6):
  - GSK Investigational Site, Bonheiden
  - GSK Investigational Site, Edegem
  - GSK Investigational Site, Ghent
  - GSK Investigational Site, Kortrijk
  - GSK Investigational Site, Leuven
  - GSK Investigational Site, Roeselare
- Bulgaria (3):
  - GSK Investigational Site, Plovdiv
  - GSK Investigational Site, Sofia
  - GSK Investigational Site, Varna
- Canada (2):
  - GSK Investigational Site, Kingston, Ontario
  - GSK Investigational Site, London, Ontario
- GSK Investigational Site, Viña del Mar, Chile
- Czechia (5):
  - GSK Investigational Site, Hradec Králové
  - GSK Investigational Site, Olomouc
  - GSK Investigational Site, Prague
  - GSK Investigational Site, Teplice
  - GSK Investigational Site, Ústí nad Orlicí
- Denmark (4):
  - GSK Investigational Site, Aalborg
  - GSK Investigational Site, Aarhus
  - GSK Investigational Site, Herlev
  - GSK Investigational Site, Koebenhavn NV
- Estonia (2):
  - GSK Investigational Site, Tallinn
  - GSK Investigational Site, Tartu
- France (4):
  - GSK Investigational Site, Clichy
  - GSK Investigational Site, Lille
  - GSK Investigational Site, Paris
  - GSK Investigational Site, Saint-Priest-en-Jarez
- Germany (16):
  - GSK Investigational Site, Heidelberg, Baden-Wurttemberg
  - GSK Investigational Site, Mannheim, Baden-Wurttemberg
  - GSK Investigational Site, Ulm, Baden-Wurttemberg
  - GSK Investigational Site, Weiden, Bavaria
  - GSK Investigational Site, Frankfurt am Main, Hesse
  - GSK Investigational Site, Brinkum/Stuhr, Lower Saxony
  - GSK Investigational Site, Hanover, Lower Saxony
  - GSK Investigational Site, Rostock, Mecklenburg-Vorpommern
  - GSK Investigational Site, Cologne, North Rhine-Westphalia
  - GSK Investigational Site, Minden, North Rhine-Westphalia
  - GSK Investigational Site, Dresden, Saxony
  - GSK Investigational Site, Halle, Saxony-Anhalt
  - GSK Investigational Site, Magdeburg, Saxony-Anhalt
  - GSK Investigational Site, Jena, Thuringia
  - GSK Investigational Site, Berlin
  - GSK Investigational Site, Hamburg
- Greece (3):
  - GSK Investigational Site, Athens
  - GSK Investigational Site, Heraklion, Crete
  - GSK Investigational Site, Ioannina
- Hong Kong (2):
  - GSK Investigational Site, Hong Kong
  - GSK Investigational Site, Shatin, New Territories
- Hungary (6):
  - GSK Investigational Site, Békéscsaba
  - GSK Investigational Site, Budapest
  - GSK Investigational Site, Debrecen
  - GSK Investigational Site, Mosonmagyaróvár
  - GSK Investigational Site, Szekszárd
  - GSK Investigational Site, Vác
- Israel (10):
  - GSK Investigational Site, Afula
  - GSK Investigational Site, Beersheba
  - GSK Investigational Site, Haifa
  - GSK Investigational Site, Holon
  - GSK Investigational Site, Jerusalem
  - GSK Investigational Site, Kfar Saba
  - GSK Investigational Site, Petah Tikva
  - GSK Investigational Site, Ramat Gan
  - GSK Investigational Site, Tel Aviv
  - GSK Investigational Site, Ẕerifin
- GSK Investigational Site, Genova, Italy
- Japan (11):
  - GSK Investigational Site, Aichi
  - GSK Investigational Site, Fukuoka
  - GSK Investigational Site, Hiroshima
  - GSK Investigational Site, Hokkaido
  - GSK Investigational Site, Hyōgo
  - GSK Investigational Site, Kagoshima
  - GSK Investigational Site, Kanagawa
  - GSK Investigational Site, Osaka
  - GSK Investigational Site, Shizuoka
  - GSK Investigational Site, Tokyo
  - GSK Investigational Site, Wakayama
- Netherlands (4):
  - GSK Investigational Site, Amsterdam
  - GSK Investigational Site, Ede
  - GSK Investigational Site, Eindhoven
  - GSK Investigational Site, Rotterdam
- New Zealand (7):
  - GSK Investigational Site, Canterbury
  - GSK Investigational Site, Dunedin
  - GSK Investigational Site, Hamilton
  - GSK Investigational Site, Lower Hutt
  - GSK Investigational Site, Otahuhu
  - GSK Investigational Site, Takapuna, Auckland
  - GSK Investigational Site, Tauranga
- Poland (4):
  - GSK Investigational Site, Bydgoszcz
  - GSK Investigational Site, Lublin
  - GSK Investigational Site, Sopot
  - GSK Investigational Site, Wroclaw
- Portugal (3):
  - GSK Investigational Site, Lisbon
  - GSK Investigational Site, Porto
  - GSK Investigational Site, Viseu
- Russia (9):
  - GSK Investigational Site, Irkutsk
  - GSK Investigational Site, Kazan'
  - GSK Investigational Site, Lipetsk
  - GSK Investigational Site, Moscow
  - GSK Investigational Site, Nizhny Novgorod
  - GSK Investigational Site, Rostov-on-Don
  - GSK Investigational Site, Saint Petersburg
  - GSK Investigational Site, Samara
  - GSK Investigational Site, Tomsk
- Slovakia (5):
  - GSK Investigational Site, Bratislava
  - GSK Investigational Site, Nitra
  - GSK Investigational Site, Nové Mesto nad Váhom
  - GSK Investigational Site, Prešov
  - GSK Investigational Site, Trnava
- South Korea (4):
  - GSK Investigational Site, Daegu
  - GSK Investigational Site, Pusan
  - GSK Investigational Site, Seoul
  - GSK Investigational Site, Wŏnju
- Spain (8):
  - GSK Investigational Site, Badalona
  - GSK Investigational Site, Elche
  - GSK Investigational Site, Fuenlabrada (Madrid)
  - GSK Investigational Site, Galdakao/Vizcaya
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Marbella
  - GSK Investigational Site, Sabadell (Barcelona)
  - GSK Investigational Site, Santander
- Switzerland (2):
  - GSK Investigational Site, Bern
  - GSK Investigational Site, Zurich
- Taiwan (3):
  - GSK Investigational Site, Taichung
  - GSK Investigational Site, Taipei
  - GSK Investigational Site, Taoyuan District
- GSK Investigational Site, Ankara, Turkey (Türkiye)
- Ukraine (8):
  - GSK Investigational Site, Chernivtsi
  - GSK Investigational Site, Dnipropetrovsk
  - GSK Investigational Site, Donetsk
  - GSK Investigational Site, Kharkiv
  - GSK Investigational Site, Kyiv
  - GSK Investigational Site, Odesa
  - GSK Investigational Site, Simferopol
  - GSK Investigational Site, Vinnytsia
- United Kingdom (9):
  - GSK Investigational Site, Glasgow, Lanarkshire
  - GSK Investigational Site, Harrow, Middlesex
  - GSK Investigational Site, Birmingham
  - GSK Investigational Site, Dundee
  - GSK Investigational Site, Edinburgh
  - GSK Investigational Site, London
  - GSK Investigational Site, Manchester
  - GSK Investigational Site, Newcastle upon Tyne
  - GSK Investigational Site, Oxford

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 253 participants, having moderate-to-severe Active Crohn's Disease were randomized to the study. The study was conducted from 11 November 2011 to 17 October 2013, at 113 centers in 26 countries with sites in North America, Europe, Israel, Japan, Republic of Korea, Hong Kong, Taiwan, Australia and New Zealand.
Groups:
- GSK1605786A, 500 Milligram (mg), Once Daily: Eligible participants in this arm received GSK1605786A 500 mg, once daily (two 250 mg capsules in the morning) , orally within 30 minutes of meals, for a period of 12 weeks.
- GSK1605786A, 500 mg Twice Daily: Eligible participants in this arm received GSK1605786A 500 mg twice daily (one 250 mg capsule in the morning and one 250 mg capsule in the evening), orally within 30 minutes of meals for a period of 12 weeks.
Period: Overall Study
Arm/Group | GSK1605786A, 500 Milligram (mg), Once Daily | GSK1605786A, 500 mg Twice Daily
Started | 127 | 126
Completed | 58 | 60
Not Completed | 69 | 66
Not completed — Protocol Violation | 2 | 3
Not completed — Physician Decision | 1 | 3
Not completed — Study closed/terminated | 41 | 37
Not completed — Lack of Efficacy | 10 | 16
Not completed — Adverse Event | 9 | 4
Not completed — Met Liver Chemistry Stopping criteria | 1 | 0
Not completed — Withdrawal by Subject | 5 | 3

BASELINE CHARACTERISTICS:
Groups:
- GSK1605786A 500 mg, Once Daily: Eligible participants in this arm received GSK1605786A 500 mg, once daily (two 250 mg capsules in the morning) , orally within 30 minutes of meals, for a period of 12 weeks.
- GSK1605786A 500 mg, Twice Daily: Eligible participants in this arm received GSK1605786A 500 mg twice daily (one 250 mg capsule in the morning and one 250 mg capsule in the evening), orally within 30 minutes of meals for a period of 12 weeks.
- Total: Total of all reporting groups
Arm/Group | GSK1605786A 500 mg, Once Daily | GSK1605786A 500 mg, Twice Daily | Total
Number analyzed (Participants) | 127 | 126 | 253
Age, Continuous [Mean (Standard Deviation); unit: Years] | 39.6 (13.11) | 38.5 (12.91) | 39.1 (13.00)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 63 | 64 | 127
  Male | 64 | 62 | 126
Race/Ethnicity, Customized [Number; unit: participants]
  White-Caucasian/European | 105 | 109 | 214
  White-Arabic/North African | 104 | 105 | 209
  Black | 1 | 4 | 5
  Asian-East | 13 | 13 | 26
  Asian-South East | 2 | 0 | 2
  Asian-Japanese | 2 | 1 | 3
  Native Hawaiian/Pacific Islander | 1 | 0 | 1
  Multiple race | 2 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving Clinical Response at Week 12
Description: Clinical response, defined as decrease in Crohn's disease activity index (CDAI) score, from Baseline value of >=100 points. Baseline defined as Week 0. CDAI is scoring system measuring disease severity with scores of >=220 to <=450 describing moderately-to-severely active population(higher score indicated severe disease). Contains 8 questions related to disease symptoms; soft tools in 7 days (weightage (Wt)as 2; abdominal pain over 7 days Wt= 5; general well being Wt= 7;Crohn's disease symptoms Wt=20; antidiarrhoeal medication used Wt=30; abdominal mass Wt=10; Anemia Wt=10; standard weight with Wt=1.Total CDAI score algorithmically derived from participants-reported above Crohn's disease symptoms and investigator recorded assessments, calculated by Interactive Voice Response System. Missing efficacy data, imputed using "no effect" imputation where missing was no response or no change in response (were non-responders). If baseline CDAI, < 100,participant was considered non-responder.
Time Frame: At Week 12
Population: The Intent-to-Treat (ITT) population comprised of all participants who have satisfied the eligibility criteria and were assigned with study medication.
Measure: Number; unit: Percentage of participants
Groups:
- GSK1605786A 500 mg,Twice Daily: Eligible participants in this arm received GSK1605786A 500 mg twice daily (one 250 mg capsule in the morning and one 250 mg capsule in the evening), orally within 30 minutes of meals for a period of 12 weeks.
Arm/Group | GSK1605786A 500 mg, Once Daily | GSK1605786A 500 mg,Twice Daily
Number analyzed (Participants) | 127 | 126
Percentage of participants | 25.2 | 33.3
Statistical Analysis 1: Comparison: GSK1605786A 500 mg, Once Daily vs GSK1605786A 500 mg,Twice Daily; Test type: Superiority or Other; Mean Difference (Final Values) = 8.1, 95% CI 2-sided [-3.0 to 19.3]

2. Secondary Outcome: Percentage of Participants Achieving Clinical Remission at Week 8, Week 12 and at Both Week 8 and Week 12
Description: Clinical remission is defined as a CDAI score of <150 points. CDAI is scoring system measuring disease severity with scores of >=220 to <=450 describing moderately-to-severely active population(higher score indicated severe disease). Contains 8 questions related to disease symptoms; soft tools in 7 days (weightage (Wt)as 2; abdominal pain over 7 days Wt= 5; general well being Wt= 7;Crohn's disease symptoms Wt=20; antidiarrhoeal medication used Wt=30; abdominal mass Wt=10; Anemia Wt=10; standard weight with Wt=1.Total CDAI score algorithmically derived from participants-reported above Crohn's disease symptoms and investigator recorded assessments, calculated by Interactive Voice Response System. Missing efficacy data, imputed using "no effect" imputation where missing was no response or no change in response (were non-responders). If the Baseline value was <150, the participant was not considered to have achieved remission.
Time Frame: Week 8 and Week 12
Population: ITT population
Measure: Number; unit: Percentage of participants
Arm/Group | GSK1605786A 500 mg, Once Daily | GSK1605786A 500 mg, Twice Daily
Number analyzed (Participants) | 127 | 126
Percentage of participants
  Week 8 | 11.8 | 14.3
  Week 12 | 11.8 | 17.5
  Both Week 8 and Week 12 | 7.9 | 10.3
Statistical Analysis 1: Comparison: GSK1605786A 500 mg, Once Daily vs GSK1605786A 500 mg, Twice Daily; CDAI score (Clinical remission), GSK1605786A, 500 mg QD Vs GSK1605786A, 500 mg BID; at Week 8; Test type: Superiority or Other; Mean Difference (Final Values) = 2.5, 95% CI 2-sided [-5.8 to 10.8]
Statistical Analysis 2: Comparison: GSK1605786A 500 mg, Once Daily vs GSK1605786A 500 mg, Twice Daily; CDAI score (Clinical remission), GSK1605786A, 500 mg QD Vs GSK1605786A, 500 mg BID; at Week 12; Test type: Superiority or Other; Median Difference (Final Values) = 5.6, 95% CI 2-sided [-3.0 to 14.3]
Statistical Analysis 3: Comparison: GSK1605786A 500 mg, Once Daily vs GSK1605786A 500 mg, Twice Daily; CDAI score (Clinical remission), GSK1605786A, 500 mg QD Vs GSK1605786A, 500 mg BID; at both Weeks 8 and 12; Test type: Superiority or Other; Mean Difference (Final Values) = 2.4, 95% CI 2-sided [-4.6 to 9.5]

3. Secondary Outcome: Percentage of Participants With a Clinical Response at Week 8 and at Both Week 8 and Week 12
Description: as for outcome 1
Time Frame: Both Week 8 and Week 12
Population: ITT population
Measure: Number; unit: Percentage of participants
Arm/Group | GSK1605786A 500 mg, Once Daily | GSK1605786A 500 mg, Twice Daily
Number analyzed (Participants) | 127 | 126
Percentage of participants
  Week 8 | 24.4 | 29.4
  Both Week 8 and Week 12 | 15.7 | 24.6
Statistical Analysis 1: Comparison: GSK1605786A 500 mg, Once Daily vs GSK1605786A 500 mg, Twice Daily; CDAI score (Clinical response), GSK1605786A, 500 mg QD Vs GSK1605786A, 500 mg BID at Week 8; Test type: Superiority or Other; Mean Difference (Final Values) = 5.0, 95% CI 2-sided [-6.0 to 15.9]
Statistical Analysis 2: Comparison: GSK1605786A 500 mg, Once Daily vs GSK1605786A 500 mg, Twice Daily; CDAI score (Clinical response), GSK1605786A, 500 mg QD Vs GSK1605786A, 500 mg BID at both Week 8 and Week 12; Test type: Superiority or Other; Mean Difference (Final Values) = 8.9, 95% CI 2-sided [-1.0 to 18.7]

4. Secondary Outcome: Change From Baseline in C-reactive Protein Concentration at Weeks 4, 8, and 12
Description: Blood samples were planned to be collected for the measurement of C-reactive protein at Baseline (Screening) and at Weeks 4, 8, and 12. Baseline is defined as the measurement at Screening (Day -21 to Day -1). Change from Baseline was calculated as the value at the post-Baseline time points (Week 4, week 8 and week 12) minus the value at Baseline respectively. The study was terminated prematurely due to absence of favorable benefit-to-risk profile of GSK1605786A, and thus data for this outcome measure was not collected.
Time Frame: Baseline (Screening) and Weeks 4, 8, and Week 12
Population: ITT Population.
Arm/Group | GSK1605786A 500 mg, Once Daily | GSK1605786A 500 mg, Twice Daily
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Change From Baseline in Faecal Calprotectin at Week 12
Description: Stool samples were planned to be collected for the measurement faecal calprotectin level at Baseline (Screening) and Week 12. Baseline is defined as the measurement at Screening (Day -21 to Day -1). Change from Baseline was calculated as the value at the post-Baseline time point minus the value at Baseline. The study was terminated prematurely due to absence of favorable benefit-to-risk profile of GSK1605786A, and thus data for this outcome measure was not collected.
Time Frame: Baseline (Screening) and Week 12
Population: ITT Population.
Arm/Group | GSK1605786A 500 mg, Once Daily | GSK1605786A 500 mg, Twice Daily
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Pharmacokinetics (PK) of GSK1605786A
Description: The PK analyses was planned to perform to characterize the PK of the study drug GSK1605786A, in the participant population. PK is defined as the concentration of drug in a participant's blood at certain time points after the drug was taken by mouth. PK sampling was to be conducted at week 2, 4, 6 ,8, 10 and week 12 (pre-dose, post-dose 0.5 hour (hr) to 2 hr, 3 to 6 hr, and 6 to 28 hr post-dose. The study was terminated prematurely due to absence of favorable benefit-to-risk profile of GSK1605786A, and thus the data for this outcome measure was not collected.
Time Frame: Baseline (Screening) and Week 12
Population: The PK population consisted of the participants having received investigational product (i.e., participants in the Safety population) and for whom a sample was obtained and analyzed.
Arm/Group | GSK1605786A 500 mg, Once Daily | GSK1605786A 500 mg, Twice Daily
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Pharmacogenetic Analyses
Description: Sample for the pharmacogenetic analyses was collected during any one of the Treatment Phase visit (Week 2, 4, 6, or 8 ). The pharmacogenetic analyses was planned to perform to investigate the relationship between the genetic markers with the safety and efficacy response to GSK1605786A. These pharmacogenetic analyses was not conducted following the early termination of the study. The study was terminated prematurely due to absence of favorable benefit-to-risk profile of GSK1605786A, and thus data was not collected for this outcome measure.
Time Frame: Post randomization any time during early two weeks
Population: ITT population.
Arm/Group | GSK1605786A 500 mg, Once Daily | GSK1605786A 500 mg, Twice Daily
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) and serious adverse events (SAEs) were collected from start of study treatment (Week 0) and until week 16 for participants not entering the maintenance study CCX114157, on completion of Week 12, or until final follow-up contact.
Description: SAEs and non-serious AEs were collected in participants of the Safety Population, comprised of all participants in the ITT population except those who did not received at least one dose of treatment
Arm/Group | GSK1605786A 500 mg, Once Daily | GSK1605786A 500 mg, Twice Daily
All-Cause Mortality (participants affected / at risk) | 0/127 | 0/126
Serious Adverse Events (participants affected / at risk) | 8/127 | 6/126
Other Adverse Events (participants affected / at risk) | 61/127 | 57/126
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | GSK1605786A 500 mg, Once Daily (N=127) | GSK1605786A 500 mg, Twice Daily (N=126)
Anal abscess (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 0 | 1
Tonsillitis (Infections and infestations) | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0
Cardiac failure (Cardiac disorders) | 0 | 1
Crohn's disease (Gastrointestinal disorders) | 1 | 1
Oesophageal ulcer (Gastrointestinal disorders) | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Hepatic enzyme increased (Investigations) | 1 | 0
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | GSK1605786A 500 mg, Once Daily (N=127) | GSK1605786A 500 mg, Twice Daily (N=126)
Abdominal pain (Gastrointestinal disorders) | 13 | 12
Dyspepsia (Gastrointestinal disorders) | 6 | 10
Crohn's disease (Gastrointestinal disorders) | 7 | 8
Nausea (Gastrointestinal disorders) | 9 | 5
Nasopharyngitis (Infections and infestations) | 8 | 5
Headache (Nervous system disorders) | 10 | 14
Pyrexia (General disorders) | 8 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.